CLINICAL TRIAL: NCT00932100
Title: A Study Assessing the REG1 Anticoagulation System Compared Heparin in Subjects With Acute Coronary Syndrome
Acronym: RADAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regado Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REG-CLIN211
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: ACS; Acute Coronary Syndrome; Catheterization
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Heparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- REG1-a (Experimental): Fixed dose of RB006 (anticoagulant) Variable blinded dose of RB007 (control agent)
  Interventions: Drug: REG1
- REG1-b (Experimental): Fixed dose of RB006 (anticoagulant) Variable blinded dose of RB007 (control agent)
  Interventions: Drug: REG1
- REG1-c (Experimental): Fixed dose of RB006 (anticoagulant) Variable blinded dose of RB007 (control agent)
  Interventions: Drug: REG1
- REG1-d (Experimental): Fixed dose of RB006 (anticoagulant) Variable blinded dose of RB007 (control agent)
  Interventions: Drug: REG1
- Heparin (Active Comparator): Heparin per standard of care at the local institution
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: REG1 — IV form, bolus dose. May be redosed. Control agent given as single re-dose at completion of intervention
  Arms: REG1-a; REG1-b; REG1-c; REG1-d
Drug: Heparin — IV dose per standard of care at the local institution
  Other Names: unfractionated heparin; low molecular weight heparin
  Arms: Heparin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the REG1 anticoagulation System in Acute Coronary Syndrome (ACS) patients undergoing cardiac catheterization.

DETAILED DESCRIPTION:
Primary Outcome Bleeding Secondary Outcome Ischemia

ELIGIBILITY:
Inclusion Criteria:

* Chest pain or other ischemic symptoms a minimum of 10 minutes in duration within 72 hours before anticipated cardiac catheterization;
* At least one of the following criteria are met:

  1. New or presumably new ST-segment depression of at least 1 mm or transient (30 minutes) ST-segment elevation of at least 1 mm in 2 contiguous leads;
  2. Elevated troponin I, T, or creatine phosphokinase-MB isoenzyme level within 24 hours of signing consent as defined by the universal MI definition
  3. Documented coronary artery disease as evidenced on prior angiography, or by prior angioplasty, bypass graft surgery, or myocardial infarction

Exclusion Criteria:

* Acute ST-segment elevation myocardial infarct
* Anticipated inability to perform angiography within 24 hours of dosing
* Evidence of clinical instability
* Contraindications to anticoagulant use
* Recent cardiac intervention
* Clinically abnormal laboratory or test findings during screening
* Subject is pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The composite incidence of major and minor bleeding | Through Day 30

CONTACTS AND LOCATIONS:
Overall Officials: John H Alexander, MD MHS FACC, Principal Investigator — Duke Clinical Research Institute
Locations (43):
- United States (26):
  - Heart Center Research LLC, Huntsville, Alabama
  - Mercy Heart & Vascular Institute, Sacramento, California
  - Sutter Medical Center - Sacramento, Sacramento, California
  - Scripps Mercy Hospital, San Diego, California
  - Heart & Vascular Institute of Florida, Clearwater, Florida
  - Jim Moran Heart & Vascular Research Institute, Fort Lauderdale, Florida
  - University of Florida-Medicine Cardiology Research, Gainsville, Florida
  - University of Florida at Jacksonville, Jacksonville, Florida
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - St. Luke's Idaho Cardiology Associates, Boise, Idaho
  - St. Luke's Idaho Cardiology Associates, Meridian, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The Care Group LLC, Indianapolis, Indiana
  - Cardiovascular Institute of the South - Houma, Houma, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Henry Ford Health Systems, Detroit, Michigan
  - Buffalo Heart Group, Buffalo, New York
  - University of North Carolina - School of Medicine, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Black Hills Clinical Research Center, Rapid City, South Dakota
  - North Cypress Medical Center, Cypress, Texas
  - Swedish Medical Center - Cardiovascular, Seattle, Washington
  - Heart Clinics Northwest, Spokane, Washington
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- Canada (3):
  - Vancouver Hospital, Vancouver, British Columbia
  - Hamilton Health Science, Hamilton, Ontario
  - Montreal Heart Institute Research Center, Montreal, Quebec
- Nouvelles Cliniques Nantaises, Nantes, France
- Germany (13):
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Kardiologische Praxis, Bad Soden
  - MVZ am Kuechwald GmbH Ambulantes Herzzentrum, Chemnitz
  - Klinikum Coburg GmbH 2. Med. Klinik Ebene 3 Studienbuero, Coburg
  - Universitatsklinikum Freiburg Abt. Innere Medizin III, Freiburg im Breisgau
  - Klinikum Fulda gAG Medizinische Klinik I, Fulda
  - Universitaetsklinikum Halle/Saale Klinik fÃ¼r Innere Medizin III, Halle
  - UniversitÃ¤tsklinikum Schleswig-Holstein Kiel, Kiel
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Universitaetsklinik Magdeburg Klinik fÃ¼r Kardiologie Angiologie und Pneumologie, Magdeburg
  - Carl-von-Basedow Klinikum, Merseburg
  - Klinikum der Universitaet Muenchen GroÃŸhadern Medizinische Klinik und Poliklinik I der LMU, München
  - Klinikum Quedlinburg GmbH Klinik fuer Innere Medizin und Kardiologie, Quedlinburg

REFERENCES:
- [Result] TCT-176: Access and non-Access Site Bleeding in Acute Coronary Syndrome Patients Treated with a Novel Actively Reversible Factor IXa Inhibitor. Results from the RADAR Trial J Am Coll Cardiol 2011 58: B47
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581
- [Derived] Povsic TJ, Vavalle JP, Alexander JH, Aberle LH, Zelenkofske SL, Becker RC, Buller CE, Cohen MG, Cornel JH, Kasprzak JD, Montalescot G, Fail PS, Sarembock IJ, Mehran R; RADAR Investigators. Use of the REG1 anticoagulation system in patients with acute coronary syndromes undergoing percutaneous coronary intervention: results from the phase II RADAR-PCI study. EuroIntervention. 2014 Aug;10(4):431-8. doi: 10.4244/EIJY14M06_01. PMID 24929350
- [Derived] Povsic TJ, Cohen MG, Chan MY, Zelenkofske SL, Wargin WA, Harrington RA, Alexander JH, Rusconi CP, Becker RC. Dose selection for a direct and selective factor IXa inhibitor and its complementary reversal agent: translating pharmacokinetic and pharmacodynamic properties of the REG1 system to clinical trial design. J Thromb Thrombolysis. 2011 Jul;32(1):21-31. doi: 10.1007/s11239-011-0588-3. PMID 21503856
- [Derived] Povsic TJ, Cohen MG, Mehran R, Buller CE, Bode C, Cornel JH, Kasprzak JD, Montalescot G, Joseph D, Wargin WA, Rusconi CP, Zelenkofske SL, Becker RC, Alexander JH. A randomized, partially blinded, multicenter, active-controlled, dose-ranging study assessing the safety, efficacy, and pharmacodynamics of the REG1 anticoagulation system in patients with acute coronary syndromes: design and rationale of the RADAR Phase IIb trial. Am Heart J. 2011 Feb;161(2):261-268.e1-2. doi: 10.1016/j.ahj.2010.10.022. PMID 21315207